CLINICAL TRIAL: NCT07344350
Title: A Non-randomised, Non-inferiority Comparative Study of Oral Actiskenan (Morphine Sulfate) Versus Intranasal Sufentanil in the Early Management of Severe Acute Pain in Emergency Departments.
Acronym: SA-URGE
Status: Not yet recruiting | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1455; 2025-A02437-42 (Other: ANSM register)
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Severe Acute Pain
Keywords: Emergency department; Analgesia; Actiskenan; Sufentanil; Morphine
MeSH Terms: conditions — Acute Pain; Emergencies; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intranasal sufentanil: Patients admitted to the emergency department of Emile Muller Hospital in Mulhouse, France with a score of 6 or higher on the numerical pain rating scale.
  Interventions: Drug: Intranasal Sufentanil
- Oral actiskenan: Patients admitted to the emergency departments of Sélestat Hospital, France, with a score of 6 or higher on the numerical pain rating scale.
  Interventions: Drug: Oral Actiskenan

INTERVENTIONS:
Drug: Intranasal Sufentanil — The patient receives intranasal sufentanil with an initial dose of 0.30 µg/kg, followed by a second half-dose (0.15 µg/kg) after 10 minutes. If pain relief is inadequate, additional doses may be administered at 15-minute intervals. Sufentanil is combined with oral or slow intravenous paracetamol.
  Groups: Intranasal sufentanil
Drug: Oral Actiskenan — A 10-mg oral tablet of Actiskenan is administered, in combination with paracetamol. The dose is reduced to 5 mg in patients aged over 85 years.
  Groups: Oral actiskenan

SUMMARY:
The main objective of this study is to evaluate whether the analgesic protocol combining oral Actiskenan is non-inferior to the protocol combining intranasal Sufentanil for treating severe pain in patients admitted to the emergency department.

The primary endpoint will be the difference between the numerical pain rating scale score at the initial assessment performed by the triage nurse (baseline) and the numerical pain rating scale score measured 30 minutes after treatment administration.

DETAILED DESCRIPTION:
Secondary Objectives:

1. To evaluate the non-inferiority of the analgesia protocol combining oral actiskenan compared with the protocol combining intranasal sufentanil, 60 minutes after the initial assessment.
2. To describe the adverse effects associated with the analgesia protocols. These will be recorded following initiation of the analgesia protocol and will include nausea/vomiting, respiratory depression, dizziness, and impaired alertness.

Research conduct:

The study will not affect the care provided to patients admitted to the emergency departments of the participating centres. Each department will implement its own pain management protocol in accordance with usual care at that centre (i.e., analgesic protocol combining intranasal sufentanil and paracetamol at Emile Muller Hospital - Mulhouse, France; analgesic protocol combining oral actiskenan and paracetamol at Sélestat Hospital Center).

Digital pain assessments and monitoring of treatment-related adverse effects are already part of routine clinical practice for medical and nursing staff. To collect standardized data on pain assessment and treatment-related adverse effects, medical and nursing staff will complete a data collection form for each patient included in the study.

Patient Information: An information sheet will be provided to each eligible patient upon admission. Data will be collected using the data collection form only if the patient does not object.

Data Collected: Upon admission, and subsequently at 30- and 60-minute intervals, data will be collected on the organizational context (number of patients present in the department and number of admissions per hour), patient characteristics, type of pain (medical or traumatic), concomitant medications received (including morphine titration, analgesics, and anxiolytics), and treatment tolerance (adverse effects).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with severe acute pain of medical or traumatic origin at admission, with a score of 6 or higher on the numerical pain rating scale;
* Aged 18 years or older;
* No prior use of WHO step III analgesic before admission;
* Hemodynamic, respiratory, and neurological stability;
* Patient informed about the study and not opposed to participation.

Non-Inclusion Criteria:

* Pain related to exacerbation of chronic and/or neuropathic pain;
* Sickle cell crisis;
* Patient with substance abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the emergency departments of Emile Muller Hospital in Mulhouse, France and Sélestat Hospital, France, with a score of 6 or higher on the numerical pain rating scale.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain rating scale score 30 minutes after analgesic treatment is given | 30 minutes after analgesic treatment is given
  The primary endpoint will be the difference between the numerical pain rating scale score at the initial assessment performed by the triage nurse (baseline) and the numerical pain rating scale score measured 30 minutes after treatment administration.

SECONDARY OUTCOMES:
Numerical Pain rating scale score 60 minutes after analgesic treatment is given | 60 minutes after analgesic treatment is given
  The primary endpoint will be the difference between the numerical pain rating scale score at the initial assessment performed by the triage nurse (baseline) and the numerical pain rating scale score measured 60 minutes after treatment administration.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Sélestat, Sélestat, Bas-Rhin
  - Hôpital Emile Muller, Mulhouse, Haut-Rhin

IPD SHARING:
Plan to Share IPD: No